CLINICAL TRIAL: NCT01603030
Title: Efficacy of Moxifloxacin 0.5%/Prednisolone 1% Fixed Combination Compared With Individual Administration of Moxifloxacin 0.5% and Prednisolone 1% in the Prevention of Post Operative Inflammation in Patients Having Lasik Surgery
Brief Title: Efficacy of Moxifloxacin/Prednisolone in Prevention of Post Surgery Inflammation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Adapt Produtos Oftalmológicos Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADAMOXPRE01/10
Record Dates: First submitted 2011-03-22; First posted 2012-05-22 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Eye Infection/Inflammation Other
Keywords: Moxifloxacin; Prednisolone; LASIK
MeSH Terms: conditions — Eye Infections | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- moxifloxacin/prednisolone combination (Experimental): 1 gtt, 4x/day, 15 days
  Interventions: Drug: moxifloxacin/prednisolone combination
- moxifloxacin 0,5% + Prednisolone 1% (Active Comparator): 1 drop of each bottle, BID, 15 days
  Interventions: Drug: moxifloxacin 0,5% + prednisolone 1%

INTERVENTIONS:
Drug: moxifloxacin 0,5% + prednisolone 1% — 1 gtt, 4x/day, 15 days
  Other Names: moxifloxacin 0,5%, prednisolone 1%
  Arms: moxifloxacin 0,5% + Prednisolone 1%
Drug: moxifloxacin/prednisolone combination — 1 gtt, 4x/day, 15 days
  Other Names: moxifloxacin 0,5%; predfort
  Arms: moxifloxacin/prednisolone combination

SUMMARY:
This is a Unicentric, double-blind, randomized, two-arm, parallel-group study to demonstrate the efficacy of moxifloxacin/prednisolone acetate fixed combination compared with individual administration of moxifloxacin + acetate Prednisolone Eye drops in Prevention of Post Operative Inflammation and Infection in LASIK surgery.

DETAILED DESCRIPTION:
antibiotic/steroid combination compared to individuals components 15 days of treatment

ELIGIBILITY:
Inclusion Criteria:

* Men or women of any race, between 18 and 50 years of age up to 8 degrees of myopia or hyperopia of up to 04 degrees or up to 3 degrees without astigmatism and other eye problems associated.
* Able to understand and provide informed consent,
* Willingness to complete all required study visits,
* Willingness to undergo surgery to correct grade (myopia, astigmatism, hyperopia) by LASIK in both eyes (at the same surgical or surgical procedures separated) or in only one eye.
* Examination of normal fundus by direct ophthalmoscopy or indirect;
* Measurements of intraocular pressure (IOP), treated or untreated, less than or equal to 20 mmHg. Individuals with glaucoma / ocular hypertension are eligible if their blood pressure is controlled by a single ocular hypotensive agent with the exception noted in criterion of exclusion. 16.
* Women who may become pregnant (those that are not surgically sterile or postmenopausal) may participate in the study if they meet all the following conditions: a)not breastfeeding; b)have a negative pregnancy test at screening prior to recruitment; c)agree to submit to a urine test for pregnancy at the time of its withdrawal from the study; d)not to conceive during the study period; e)are using birth control methods appropriate and agrees to continue to use birth control methods appropriate for the duration of the study (the methods of birth control are adequate: hormonal contraceptives - oral, implantable or injectable; mechanics - spermicide associated with a barrier method like a condom or diaphragm, IUD, or sterilization of the partner).

Exclusion Criteria:

* Glaucoma or intraocular hypertension not controlled;
* Use of nonsteroidal antiinflammatory drugs (NSAIDs) ocular topical or systemic drugs (NSAIDs) during the study and the 14 days prior to study entry, except for an allowed daily dose of aspirin low-dose (100 mg);
* Ocular anti-infective drug use during the study and within 30 days prior to study entry or any other eye medicines with the exception noted in criterion Insertion 6.
* Topical steroids, inhaled or systemic ocular during the study and the 14 days prior to study entry;
* Ocular trauma in the eye prior to operate (including intraocular surgery in the previous twelve months due to trauma or cataract in the past);
* History of chronic ocular inflammatory disease or recurrent (ie, iritis, scleritis, uveitis, iridocyclitis, rubeosis iridis) in the eye to be operated;
* Any intraocular inflammation (score of cells than Grade 0) to be present during the examination of slit lamp or ocular pain increased in the Grade 1 -2 Day in the study eye (eye operation);
* Proliferative diabetic retinopathy (eye operation) non-proliferative diabetic retinopathy, moderate to severe (eye operation);
* Uncontrolled diabetes mellitus;
* Patients with vision in one eye or vision not correctable to LogMAR 1.0 or better in each eye using the ETDRS framework;
* Participation in any other clinical study within 12 months prior to surgery, pregnant women, lactating or under conditions of breeding methods that are not using adequate birth control (as defined in the criteria for inclusion, above);
* Known or suspected allergy or hypersensitivity to moxifloxacin, steroids, topical anesthetics or any other component of the study medication;
* History or other evidence of severe illness, or other systemic conditions that may cause the patient, in the opinion of the Investigator, the study is inadequate;
* Patients with epithelial herpes simplex (dendritic keratitis), vaccinia, varicella, or other viral disease of the cornea or conjunctiva, tuberculosis of the eye, fungal diseases of ocular structures;
* Patients who use a topical ophthalmic prostaglandin, such as ,Travatan® (travoprost),Xalatan®(latanoprost),Lumigan®(bimatoprost)and Rescula®(unoprostone) should discontinue their use starting four days before surgery until their departure from study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-08 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Day 15 Evaluation of Anterior Chamber | 15 days
  The primary efficacy variable of this study is the percentage of patients with a score of zero postoperative inflammation (anterior chamber inflammation, ie, presence of cells in the anterior chamber (0-4) in the study on Day 15. The absence of bacterial infection on Day 15 ± 1 will be assumed to demonstrate that the antibacterial agents in the association of moxifloxacin / acetate Prednisolona1% and moxifloxacin + acetate Prednisolona1% Eye drops are equal in antimicrobial effectiveness, and that they acted in a prophylactic manner to prevent of bacterial infection.

SECONDARY OUTCOMES:
day 15 physician´s follow-up impression of inflammatory reaction score | 15 days
  the clinical evaluation will be based on the following variables: IOP, assessment of visual acuity, slit lamp examination (lids, conjunctiva, cornea), and examination of the fundus (retina / macula / choroid, vitreous and optic nerve).

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Mucioli, Dra., Study Chair — Universidade Federal de São Paulo - Hospital São Paulo - UNIFESP
Locations (1):
- Universidade Federal de São Paulo - Hospital São Paulo - UNIFESP, São Paulo, SP/Brazil, Brazil